CLINICAL TRIAL: NCT06615778
Title: Effectiveness of Motivated Social Motional Learning (MSEL) on Bullying Among Hong Kong Primary School Students: a Three-Arm Cluster Randomized Control Trial
Brief Title: Effectiveness of Motivated Social Motional Learning (MSEL) Program on Bullying Among Hong Kong Primary School Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr.Yik-Wa Law, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA230558
Record Dates: First submitted 2024-09-15; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Bullying of Child
Keywords: Bullying perpetration and victimization

STUDY DESIGN:
Masking Description: Due to the nature of the RCT, blinding the trial participants, school officials, and teachers is not possible. Also, the investigator and the outcome assessor cannot be masked in the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Waitlist Control Group (No Intervention): The waitlist control arm consists of participants who are randomly assigned to not receive any treatment. This group will continue with their regular school curriculum and activities, without any additional programming or modifications. The purpose of the control group is to provide a point of comparison for the outcomes measured in the two experimental groups that receive different intervention. If the study shows that the intervention is effective, they will receive all the intervention components of MSEL the in following school year.
- Curriculum-based Social-Emotional Learning (CSEL) (Experimental): 6-session SEL training will be delivered as the experimental component in this arm. The primary goal of the SEL training is to reduce bullying and cyberbullying perpetration and victimization by enhancing students' social-emotional competence, which has been examined to be the protective factor for bullying-related behaviors (Espejo-Siles et al., 2020; Zych et al., 2018). Additionally, due to the interactive and cooperative nature of the SEL curriculum, it is also beneficial for improving interpersonal relatedness (i.e., peer relationships, teacher-student relationships) within the class, which according to past research, is also associated with reduced bullying behaviors (Durlak, Mahoney, & Boyle, 2022). Each session lasts 40 minutes and will be delivered by the headteacher who will received systematic training on SEL instructions in each class.
  Interventions: Behavioral: Curriculum-based Social Emotional Learning
- Motivated Social Emotional Learning (Experimental): MSEL arm consists of three intervention components: 1) CSEL, 2) the Class Ambassador (meaningful role-taking), and 3) Secret Angel . Participants in this arm will receive the same 6-session SEL training as participants in the CSEL arm. Other than CSEL, the second component is the Class Ambassador, adapted from the pupil responsibilities intervention developed by Ellies et al. (2016). The main goal of Class Ambassador is to offer autonomous, prosocial ways of acquiring recognition and social status through a variety of daily classroom jobs. The objective of Class Ambassador is to provide opportunities for students to 1) practice their social-emotional skills, 2) establish healthy peer relationships, 3) autonomously performing prosocial roles and fulfilling social responsibilities. The third component is the Secret Angel. Students will be observe, record, recognize each other's performance anonymously through appraisal notes.
  Interventions: Behavioral: Motivated Social Emotional Learning

INTERVENTIONS:
Behavioral: Motivated Social Emotional Learning — MSEL arm consists of three intervention components: 1) CSEL, 2) the meaningful role tasks, and 3) the Secret Angel activity. First, participants in the MSEL arm will receive the same 6-session SEL as participants in the Curriculum-based Social-Emotional Learning arm.
  Second, other than the CSEL, the second component is the Class Diploma tasks adopted from the pupil responsibilities intervention developed by Ellies et al. (2016). Participants will be provided with a list of meaningful roles and select the role they are willing to take based on their talents and interests. Each participant will take the role for two weeks, fulfilling the related duties and responsibilities. The third component is the Secret Angel, in which participants will anonymously recognize each other via the appraisal notes on Shout Out for Your Board.
  Arms: Motivated Social Emotional Learning
Behavioral: Curriculum-based Social Emotional Learning — In the CSEL arm, 6-session SEL training will be delivered as the experimental component. The primary goal of the SEL training is to reduce traditional bullying and cyberbullying perpetration and victimization by enhancing students' social-emotional competence, which has been examined to be the protective factor for bullying-related behaviors.
  Each session lasts 40 minutes and is delivered by the headteacher in each class weekly as an after-school workshop. The SEL curriculum is tailored to the social-emotional needs of primary school students, as suggested by CASEL (2013). Also, building on past literature highlighting the lack of SEC as a risk factor linked to bullying behaviors both in the physical and cyber world, specific topics such as self-appreciation (self-awareness), stress management (self-management), respect and acceptance (social awareness), and conflict resolution (relationship skills) incorporated into the curriculum design.
  Arms: Curriculum-based Social-Emotional Learning (CSEL)

SUMMARY:
The present study aimed to test the effectiveness of motivated social-emotional Learning (MSEL) and traditional curriculum-based social-emotional learning (CSEL) in reducing bullying perpetration and victimization among Hong Kong primary school students. The main research questions the cRCT aims to answer are:

1. Does MSEL reduce bullying perpetration and victimization among Hong Kong primary school students?
2. Is MSEL more effective than the traditional CSEL in reducing bullying perpetration and victimization among Hong Kong primary school students?

In according with the research questions, the following hypotheses will be tested:

H1: MSEL can significantly change primary outcomes and secondary outcomes at posttest and 3-month follow-up.

H2: CSEL can significantly change primary outcomes and secondary outcomes at posttest and 3-month follow-up.

H3: Compared with the intervention group of CSEL, the MSEL group will experience greater changes in primary and secondary outcomes.

Classroom is the randomization unit and the participating classrooms are randomly assigned to each of the three arms-the waitlist control group (WCL, no intervention delivered during the implementation period), the CSEL group (only receiving curriculum-based SEL training), and the MSEL group (participating in CSEL and Class Ambassador). The multi-method (i.e., questionnaires and face-to-face interviews) approach will be used to assess primary outcomes (i.e., school bullying victimization and perpetration, cyberbullying perpetration, defending behaviors) and secondary outcomes (i.e., social-emotional competence, prosocial behaviors, school safety and liking, psychological well-being). Also, the data collection will be conducted in the 2024-2025 academic term at three different time points: the baseline (T0, prior to the beginning of intervention, Sept. 2024), the posttest (T1, the completion of intervention, Dec. 2024) and the follow-up (T2, three months after the completion of intervention, April 2025). The analysis and report of the data start in the fall of 2025.

DETAILED DESCRIPTION:
Informed by self-determination theory and the evolutionary theory, the intervention aims to enable primary school students in Hong Kong to enhance behavioral management and choose healthier behaviors by 1) promoting their autonomy, relatedness, and competence; and 2) achieving more social rewards through prosocial opportunities. These are theorized as being facilitated by 1) autonomy in taking pro-social responsibilities, 2) competence empowerment, and 3) interpersonal relatedness (teacher-student and peer relatedness). The intervention aims to do so via three intervention components (see intervention logic model Appendix Figure A1). First, social-emotional learning (SEL) will be delivered to students to improve students competence in five developmental domains (i.e., self-awareness, social-awareness, self-management, responsible decision-making, and relationship skills. Second, students will be offered the opportunity to autonomously take responsible and meaningful roles and to earn social benefits. Third, built on meaningful role-taking, students will recognize and connect to others by expressing compliments and by helping others in need in their own ways. The above three components will serve as both the universal and indicated approach. The universal approach aims at reducing misconduct and enhancing prosocial behaviors among all students. The indicated approach, through the use of tailored social roles and application of SEL training with specific topics (e.g., stress management, conflict solving, interpersonal skill lab), targets socially integrated bullies and socially marginalized bullies respectively.

Schools are recruited voluntarily. Based on the inclusion criteria, all eligible schools will be identified from the list of primary schools in Hong Kong, totaling 477, obtained from the Hong Kong Education Bureau. With the support of a local NGO, invitations will be sent to all qualifying middle-band schools through the nonprofit organization. In the invitation email, schools will receive information about training, implementation, and the nature of the proposed evaluation to gain their initial interest and commitment. Participation will be offered on a first-come-first-served basis to schools that respond to the invitation email and confirm their commitment, in writing, to (1) deliver the assigned intervention program and (2) participate in the evaluation. If parents or caregivers are willing to have their children participate in the CRCT, they will be required to provide informed written consent. Meanwhile, parents can request the withdrawal of their children from the trial assessments at baseline or at any other time throughout the project. Additionally, students will sign an assent to indicate their agreement or disagreement to participate in the research.

The author of the study and the registered social workers (RSW) from the collaborated agency will coach and support the intervention schools throughout the implementation. Each facilitator (headteacher from each class) will be assigned to a supervisor (RSW) to discuss the implementation. Meanwhile, five fidelity control methods will be applied in this program.

1. Programme manuals. Detailed program manuals are tailored for different intervention components in CSEL and MSEL arms. The program manual for the CSEL group includes all the details regarding the operation of the 6-session SEL curriculum. For the MSEL group, other than the program manual for SEL curriculum, the program manuals for meaningful role-taking and secret angel are also for headteachers.
2. Intervention training. Before the intervention begins, headteachers in the intervention group will be systematically trained for 2 times (2 hours each), which fully covers the operation of program manuals. First, headteachers in CSEL will be trained in delivering the SEL curriculum. Headteachers will be provided with the opportunities to go through the manual with the trainers (professional social workers from the collaborated agency) and empowered with SEL-related techniques (e.g., ROPE for SEL training rules) and skills (e.g., cultivating a safe environment for sharing) through various training setups, such as role-play, group activities and mock class.
3. SEL lesson report. Facilitators will fill out a lesson report form each time they deliver an SEL session.
4. Implementation checklist. To verify intervention fidelity, two individuals who are not members of the program will observe the implementation of all intervention components and document the concordance between a prespecified checklist of elements for the intervention and the actual implementation itself. These checklists are developed separately for each intervention component. Interrater reliability using the Kappa statistic will be computed to assess the coding reliability.
5. Biweekly and monthly meetings. Facilitators and their assigned supervisors will conduct biweekly meetings to discuss the lesson report, teaching strategies, and other contingencies. Additionally, monthly meetings will be held between the research team and supervisors to check on the implementation of the intervention and to fix problems if necessary.

ELIGIBILITY:
* The inclusion criteria for schools, classes, and students are as follows.

  1. Primary School: To reduce the confounding effect of academic achievements on student behavior, only public schools in the middle band (i.e., the middle 33% of academic ratings) in Hong Kong will be included in the sampling. Single-sex schools will be excluded in consideration of the sampling diversity. Furthermore, schools implementing other manualized anti-bullying programs will not be included.
  2. Classes: The inclusion criteria are classes from Grade 4 and 6 (ages 9-13 years old). This research specifically targets classes in Grades 4 and 6 for several reasons. First, studying the integration of adaptive and maladaptive functions of problematic behaviors during this sensitive period may have a greater impact on young adolescents (Ellis et al., 2011). Secondly, a meta-analysis conducted by Yeager et al. (2015) reveals that the effectiveness of anti-bullying interventions declines significantly after Grade 7. Hence, the trial focuses on classes in Grades 4-6.
  3. Students: Inclusion criteria for students specify that they must be enrolled in the class and regularly attend its lessons.
* The exclusion criteria schools executing other manualized anti-bullying programs are excluded in this intervention.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Defending Behavior in bullying incidents | Baseline, 3-month and 6-month
  Defending behavior in bullying incidents is assessed with three items from the larger Bystander Behavior Scale (Jungert et al., 2016), using a 4-point Likert scale ( 1= Has not happened, 2 = Only once or twice, 3 = 2 or 3 times a month, 4= About once a week, 5 = Several times a week). Students are asked how often they defend the bullying victims in the last semester in the way of 1) comforting the victim, 2) telling others to stop bullying, and 3) trying to make others stop bullying. The total score ranges from 4 to 20, with higher scores indicating more frequent defending behaviors.
Cyberbullying Perpetration | Baseline, 3-month and 6-month
  Cyberbullying Perpetration is measured with a 7-item Cyberbullying Perpetration and Victimization Scale (CPVS). Students are asked how many times in the last semester they had engaged in various cyberbullying behaviors through online short message services via the Internet and electronic devices (e.g., emails, blogs, Messenger, Facebook). 7 items include cursing/insulting/ humiliating, threatening/intimidating, posting or sending private/embarrassing pictures without consent, making unwanted sexual remarks, spreading rumors, and spreading a computer virus. Students indicate their cyberbullying behaviors by checking one of five categories (1=has not happened, 2=only once or twice, 3- 2 or 3 times a month, 4=about once a week, 5=several times a week). The total score ranges from 7 to 35, with higher scores indicating more frequent cyberbullying behaviors.
School bullying perpetration and victimization | Baseline, 3-month and 6-month
  School bullying perpetration and victimization are evaluated using the Chinese version of the Olweus Bully/Victim Questionnaire (C-OBVQ). Students are asked about their bullying-engaged experience in the last semester. The answers to all 12 questions can be chosen from a uniform 5-point Likert scale: has not happened, only once or twice, 2-3 times a month, once a week, and several times a week. Students who reported "2-3 times per month" or more frequently have been bullied in any form were classified as victims, participants who reported "2-3 times per month" or more frequently bullied others were deemed as bullies, participants who reported bullying perpetration and victimization simultaneously for "2-3 times per month" or more frequent were labeled as bully-victims (Solberg &amp;amp;amp; Olweus, 2003). With the total scores ranging from 12 to 60 points, a higher score indicates a higher level of school bullying perpetration and victimization.

SECONDARY OUTCOMES:
Psychological Well-being | Baseline, 3-month and 6-month
  Psychological well-being is measured using the Patient Health Questionnaire-9 (PHQ-9) (Kroenke et al., 2001; Wang et al., 2014). The PHQ-9 scale has good sensitivity and specificity in detecting depression in youth, is an effective screening tool for the risk of depression among adolescents, and has been validated in Chinese adolescents (Allgaier et al., 2012; Leung et al., 2020; Richardson et al., 2010). Participants are asked how often they had experienced depressive symptoms in the past 2 weeks (e.g., feeling tired or having little energy), with response options ranging from 0 (not at all) to 3 (nearly every day). A total PHQ-9 score (range from 0 to 27) is calculated, where a higher score indicates more depressive symptoms. PHQ-9 has been validated by Tsai et al. (2014) and is frequently used among Hong Kong young children. The internal consistency in previous research ranged from 0.82 to 0.88 (Leung et al., 2020; Leung et al., 2015; Yu et al., 2010; Zhu et al., 2023).
Social Emotional Competence (SEC) | Baseline, 3-month and 6-month
  Social Emotional Competence (SEC) is assessed with the Modified Chinese version of Delaware Social and Emotional Competencies Scale-student version (DSECS-S) consists of 22 items on a 4-point Likert scale. The modified scale is designed on five domains: responsible decision-making (e.g., "I feel responsible for how I act."), social awareness (e.g., "I think about how others feel."), self-management (e.g., "I can control how I behave."), self-awareness (e.g., "I can calm myself when upset."), and social relationship (e.g., "I get along well with others."). Respondents are asked to read statements to rate how applicable it is. The total scores of DSECS-S range from 22 to 88 points, with higher scores indicating a higher level of SEC.
School well-being | Baseline, 3-month and 6-month
  School well-being is assessed using the school safety and school liking subscales of the Chinese version of the Delaware School Climate Survey-Student (C-DSCS). Students are asked if they feel safe at school(e.g., I feel safe at this school) and if they like the school(e.g., I like this school). Students respond to 7 items on a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). Total scores range from 7 to 28 points, with higher scores indicating greater school well-being. The Chinese version of the Delaware School Climate Survey-Student (C-DSCS) has been applied among Hong Kong primary school students with high internal consistency.
Prosocial behavior | Baseline, 3-month and 6-month
  Prosocial behavior is measured using a 5-item subscale from the Strength and Difficulty Questionnaire (SDQ). Students are asked about their prosocial behaviors in the form of 1) being nice to other people, 2)sharing with others, 3) being helpful if someone is hurt, upset or feeling ill, 4) being kind to younger children, 5) voluntarily helping others. Responses are recorded on a 3-point Likert scale(1 = Not True, 3 = Certainly True), with total scores ranging from 5 to 15 points. Higher total scores reflect greater levels of prosocial behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- The Boys and Girls Clubs Association of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No